CLINICAL TRIAL: NCT01826851
Title: Parasternal Intercostal Nerve Block in Post-Cardiac Surgery Patients: A Randomized, Controlled Trial of Extended-release Liposomal Bupivacaine (Exparel) Versus Placebo
Brief Title: Parasternal Nerve Block in Cardiac Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Peter A Knight (Other)
Responsible Party: Sponsor-Investigator, Peter A Knight, Professor, Cardiac Surgery, University of Rochester
Organization: University of Rochester (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: RSRB 00044181
Record Dates: First submitted 2013-03-25; First posted 2013-04-09 (Estimated); Results first posted 2018-08-01 (Actual); Last update posted 2018-08-01 (Actual); Status verified 2018-07

CONDITIONS: Coronary Artery Disease; Pain, Postoperative
Keywords: Pain management; Anesthetic, local; Nerve blockade; Coronary Artery Bypass Surgery; Analgesics, opioid; Postoperative complications; Bupivacaine
MeSH Terms: conditions — Coronary Artery Disease; Pain, Postoperative; Agnosia; Postoperative Complications

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Exparel (Experimental): 266 mg Exparel, single-dose injection.
  Interventions: Drug: Exparel
- Placebo (Placebo Comparator): 0.9% Normal saline, single-dose injection.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Exparel — Patients in this group will receive 266 mg Exparel diluted with 0.9% normal saline to a total volume of 50 mL and administered via parasternal intercostal nerve block prior to sternal closure.
  Post-operatively, patients will receive IV fentanyl as needed in the ICU while still intubated. A fentanyl PCA pump will be set up post-extubation as soon as possible and prior to the patient leaving the ICU.
  Other Names: SKY0402; Bupivacaine liposome extended-release injectable suspension
  Arms: Exparel
Drug: Placebo — Patients in this group will receive 50 mL of 0.9% normal saline as a parasternal intercostal nerve block prior to sternal closure.
  Post-surgical pain management will be the same as for the Exparel group.
  Other Names: Preservative-free normal saline
  Arms: Placebo

SUMMARY:
Exparel is a new local analgesic (numbing medication) that is intended to be longer acting than currently available local analgesics. The purpose of this study is to determine whether use of Exparel to numb the nerves along the breastbone after open heart surgery, will decrease pain and pain medication use after surgery.

DETAILED DESCRIPTION:
This is a Phase 2, single-institution, randomized, double-blind, parallel-group, placebo-controlled trial of patients undergoing a median sternotomy for primary cardiopulmonary bypass grafting (CABG) surgery.

78 subjects (39 per treatment arm) will be randomized in a 1:1 ratio to receive a single-dose, parasternal nerve block with either 266 mg Exparel or placebo (0.9% normal saline solution). The nerve blocks will be performed under direct visualization at the end of surgery, just prior to sternal closure.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 years old
* non-emergent coronary artery bypass grafting surgery (on and off pump)
* median sternotomy

Exclusion Criteria:

* Concomitant cardiac procedures (e.g. aortic valve repair/replacement, mitral valve repair/replacement, aortic root replacements).
* Redo sternotomy.
* < 50 kg (Exparel® is currently only approved in patients > 50 kg).
* Pregnant or nursing
* History of alcohol, narcotic or illicit drug abuse
* Participation in another study evaluating investigational medications within the past 30 days
* Taking narcotic analgesics within 3 days pre-operatively or perioperative stress-dose steroids.
* Chronic non-cardiac pain (e.g. lower back pain, fibromyalgia) requiring narcotic analgesics.
* Pre-operative mild liver insufficiency as defined by liver function tests [(i.e. alanine aminotransferase (ALT), aspartate aminotransferase (AST)] ≥ 1.5 times the upper limit of normal (ULN: ALT: 0-35 U/L, AST: 0-35 U/L, Alk Phos 35-105 U/L, Total bilirubin: 0-1.2 mg/dL)
* Pre-operative mild renal insufficiency (Cr ≥ 1.5 mg/dL)
* Allergy to amide-type anesthetics
* Recurrent ventricular arrhythmias, low cardiac output requiring inotrope and/or intra-aortic balloon pump support, left ventricular ejection fraction < 30% at time of pre-operative screening/evaluation.
* Unable to provide informed consent or unable to understand how to use pain rating scales.
* Inability to understand or operate the patient-controlled analgesia (PCA) machine.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 79 (Actual)
Dates: Start 2013-03; Primary Completion 2017-06 (Actual); Study Completion 2017-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Peter A Knight, MD, Principal Investigator — University of Rochester
Locations (1):
- University of Rochester Medical Center, Rochester, New York, United States

REFERENCES:
- [Derived] Lee CY, Robinson DA, Johnson CA Jr, Zhang Y, Wong J, Joshi DJ, Wu TT, Knight PA. A Randomized Controlled Trial of Liposomal Bupivacaine Parasternal Intercostal Block for Sternotomy. Ann Thorac Surg. 2019 Jan;107(1):128-134. doi: 10.1016/j.athoracsur.2018.06.081. Epub 2018 Aug 28. PMID 30170012

RESULTS

PARTICIPANT FLOW:
Groups:
- Exparel: 266 mg Exparel, single-dose injection.
  Exparel: Patients in this group will receive 266 mg Exparel diluted with 0.9% normal saline to a total volume of 50 mL and administered via parasternal intercostal nerve block prior to sternal closure.
  Post-operatively, patients will receive IV fentanyl as needed in the ICU while still intubated. A fentanyl PCA pump will be set up post-extubation as soon as possible and prior to the patient leaving the ICU.
- Placebo: 0.9% Normal saline, single-dose injection.
  Placebo: Patients in this group will receive 50 mL of 0.9% normal saline as a parasternal intercostal nerve block prior to sternal closure.
  Post-surgical pain management will be the same as for the Exparel group.
Period: Overall Study
Arm/Group | Exparel | Placebo
Started | 38 | 41
Completed | 38 | 41
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Exparel | Placebo | Total
Number analyzed (Participants) | 38 | 41 | 79
Age, Categorical [Count of Participants; unit: Participants]
  Age Distribution: <=18 years | 0 | 0 | 0
  Age Distribution: Between 18 and 65 years | 16 | 24 | 40
  Age Distribution: >=65 years | 22 | 17 | 39
Age, Continuous [Mean (Standard Deviation); unit: years] | 66 (7.7) | 64 (8.6) | 65 (8.19)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 5 | 12
  Male | 31 | 36 | 67
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 38 | 40 | 78
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 38 | 41 | 79
BMI [Mean (Standard Deviation); unit: kg/m^2] | 31 (4.8) | 30.4 (4.7) | 30.7 (4.7)

OUTCOME MEASURES:

1. Primary Outcome: Median Cumulative Morphine Equivalent
Description: The cumulative opioid requirement is reported as morphine equivalent. The total amount of narcotics required by the subjects in the Exparel group and placebo group were measured at 1,2,4,8,12,24,36,48,60, and 72 hours post-injection of Exparel or 0.9% normal saline. The amounts were analyzed and are reported as morphine equivalents.
Time Frame: Outcome was measured at 1,2,4,8,12,24,36,48,60, and 72 hours post intercostal nerve block.
Measure: Median (Inter-Quartile Range); unit: Morphine Equivalents
Arm/Group | Exparel | Placebo
Number analyzed (Participants) | 38 | 41
Morphine Equivalents
  1 hour post injection | 0 [0 to 0] | 2.5 [0 to 1.25]
  2 hours post injection | 0 [0 to 5] | 5 [0 to 5]
  4 hours post injection | 5 [0 to 5] | 8.4 [0 to 5]
  8 hours post injection | 5 [0 to 9.87] | 6 [3.5 to 15]
  12 hours post injection | 13 [1 to 11.35] | 16 [2 to 12]
  24 hours post injection | 11.5 [7 to 22.15] | 18 [10.75 to 29]
  36 hours post injection | 8.5 [3.06 to 25.37] | 15 [9 to 42]
  48 hours post injection | 4.167 [2.12 to 26.47] | 3.33 [7.5 to 21.25]
  60 hours post injection | 4.167 [0.46 to 6.67] | 3.33 [1.67 to 8.3]
  72 hours post injection | 2.5 [0 to 5] | 3.33 [0 to 6.67]

2. Primary Outcome: Median Pain Levels
Description: The pain scores of the subjects in the Exparel group and placebo group were measured at 1,2,4,8,12,24,36,48,60, and 72 hours post-injection of Exparel or 0.9% normal saline. The pain scores were reported on a scale of 0 - 10. 0 being no pain. 10 being the worst pain.
Time Frame: Outcome was measured at 1,2,4,8,12,24,36,48,60, and 72 hours post intercostal nerve block.
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Exparel | Placebo
Number analyzed (Participants) | 38 | 41
units on a scale
  1 hour post injection | 0 [0 to 0] | 0 [0 to 0]
  2 hours post injection | 0 [0 to 0] | 0 [0 to 1]
  4 hours post injection | 0 [0 to 1] | 0 [0 to 3.25]
  8 hours post injection | 0 [0 to 2.75] | 2 [0 to 5]
  12 hours post injection | 1.5 [0 to 3.75] | 2 [0 to 4]
  24 hours post injection | 2 [0 to 4] | 4 [0 to 5]
  36 hours post injection | 2 [0 to 4] | 2 [0 to 5]
  48 hours post injection | 1.5 [0 to 3.75] | 2 [0 to 4]
  60 hours post injection | 0 [0 to 2] | 0 [0 to 2]
  72 hours post injection | 1 [0 to 3] | 0 [0 to 3]

3. Secondary Outcome: Time to Extubation (Hours)
Description: Time to remove endotracheal tube following surgery.
Time Frame: 77 hours
Measure: Median (Inter-Quartile Range); unit: Hours
Arm/Group | Exparel | Placebo
Number analyzed (Participants) | 38 | 41
Hours | 6.8 [4.2 to 9.6] | 6.4 [4.3 to 10.9]

4. Secondary Outcome: ICU Length of Stay (Hours)
Description: Duration of time spent in the intensive care unit postoperatively.
Time Frame: 135 hours
Measure: Median (Inter-Quartile Range); unit: Hours
Arm/Group | Exparel | Placebo
Number analyzed (Participants) | 38 | 41
Hours | 25 [19 to 47] | 22.8 [19 to 42]

5. Secondary Outcome: Time to First Bowel Movement (Days)
Description: Time to first bowel movement following surgery.
Time Frame: 35 days
Population: Data was not collected on 3 participants in the Exparel arm and 1 participant in the Placebo arm.
Measure: Median (Inter-Quartile Range); unit: Days
Arm/Group | Exparel | Placebo
Number analyzed (Participants) | 35 | 40
Days | 2 [2 to 3] | 2 [2 to 3]

6. Secondary Outcome: Hospital Length of Stay (Days)
Description: Duration of time spent in the hospital following surgery.
Time Frame: 25 days
Measure: Median (Inter-Quartile Range); unit: Days
Arm/Group | Exparel | Placebo
Number analyzed (Participants) | 38 | 41
Days | 5 [4 to 7] | 5 [4 to 6]

7. Secondary Outcome: Time to Return to Work or Daily Activities
Description: Time to return to work or daily activities following surgery will be assessed at postoperative clinic follow up or during a follow up telephone interview.
Time Frame: 36 days
Population: Data was not collected on 15 participants in the Exparel arm and 17 participant in the Placebo arm.
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Exparel | Placebo
Number analyzed (Participants) | 23 | 24
Days | 21.8 (6.9) | 21.3 (7.7)

ADVERSE EVENTS:
Time Frame: Adverse event data were collected at throughout a 72 hour post intercostal nerve block at 1, 2, 4, 8, 12, 24, 36, 48, 60, and 72 hours. Adverse event data was also collected at the time of follow-up, which occurred at 3-4 weeks post-operatively.
Arm/Group | Exparel | Placebo
All-Cause Mortality (participants affected / at risk) | 0/38 | 0/41
Serious Adverse Events (participants affected / at risk) | 4/38 | 10/41
Other Adverse Events (participants affected / at risk) | 38/38 | 40/41
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Exparel (N=38) | Placebo (N=41)
Suspected bupivacaine toxicity (General disorders) | 0 (0) | 0 (0)
Myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0)
Transient ischemic attack (Nervous system disorders) | 0 (0) | 0 (0)
Cerebral vascular accident with permanent deficits (Nervous system disorders) | 1 (1) | 0 (0)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Sepsis (Infections and infestations) | 0 (0) | 0 (0)
Mediastinitis (Infections and infestations) | 0 (0) | 0 (0)
Sternal wound dehiscence (Surgical and medical procedures) | 0 (0) | 0 (0)
Reoperation due to graft failure (Surgical and medical procedures) | 0 (0) | 0 (0)
Reoperation for bleeding (Surgical and medical procedures) | 0 (0) | 0 (0) — Return to OR for bleeding
Renal failure requiring hemodialysis (Renal and urinary disorders) | 0 (0) | 0 (0)
Phrenic nerve Injury (Surgical and medical procedures) | 0 (0) | 0 (0)
Readmission to ICU (General disorders) | 0 (0) | 0 (0)
Deep venous thrombosis (Vascular disorders) | 0 (0) | 0 (0)
Pulmonary embolism (Vascular disorders) | 0 (0) | 0 (0)
New onset SVT or ventricular tachycardia (Cardiac disorders) | 3 (3) | 6 (6)
Heart Failure (Cardiac disorders) | 0 (0) | 0 (0)
Coma (Nervous system disorders) | 0 (0) | 0 (0)
Encephalopathy (Nervous system disorders) | 0 (0) | 0 (0)
Acute limb ischemia (Vascular disorders) | 0 (0) | 0 (0)
Multiorgan failure (General disorders) | 0 (0) | 0 (0)
Aortic dissection (Vascular disorders) | 0 (0) | 0 (0)
New onset ventricular fibrillation (Cardiac disorders) | 0 (0) | 2 (2)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Exparel (N=38) | Placebo (N=41)
Atrial Fibrillation (Cardiac disorders) | 12 (12) | 13 (13)
Bradycardia (Cardiac disorders) | 6 | 4
Bundle Branch Block (Cardiac disorders) | 9 | 8
First Degree AV Block (Cardiac disorders) | 5 | 7
Premature Atrial Contraction (Cardiac disorders) | 2 | 0
Palpitations (Cardiac disorders) | 7 | 5
Prolonged QT Interval (Cardiac disorders) | 8 | 5
Premature Ventricular Contraction (Cardiac disorders) | 11 | 11
ST Changes (Cardiac disorders) | 2 | 6 — ST segment elevation or depression on electrocardiogram
Sinus Tachycardia (Cardiac disorders) | 9 | 6
Constipation (Gastrointestinal disorders) | 16 | 20
Diarrhea (Gastrointestinal disorders) | 7 | 9
Nausea (Gastrointestinal disorders) | 24 | 18
Vomiting (Gastrointestinal disorders) | 9 | 0
Anxiety (General disorders) | 9 | 16
Blurred Vision (General disorders) | 3 | 0
Chills (General disorders) | 3 | 3
Diaphoresis (General disorders) | 14 | 14 — Excessive sweating
Dizziness/Light headedness (General disorders) | 18 | 22
Fever (General disorders) | 2 | 6
Itching (General disorders) | 3 | 0
Metallic Taste in Mouth (General disorders) | 5 | 7
Restlessness (General disorders) | 12 | 15
Generalized Weakness (Musculoskeletal and connective tissue disorders) | 17 | 18
Headache (Nervous system disorders) | 4 | 7
Miosis (Nervous system disorders) | 0 | 3 — Pupillary constriction
Parasthesias (Nervous system disorders) | 5 | 13 — Numbness
Somnolence (Nervous system disorders) | 12 | 12 — Abnormal drowsiness
Tinnitis (Nervous system disorders) | 6 | 3 — Ringing in ears
Tremors (Nervous system disorders) | 2 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-02-15): https://cdn.clinicaltrials.gov/large-docs/51/NCT01826851/Prot_SAP_000.pdf